CLINICAL TRIAL: NCT03709901
Title: Viable Allograft Supplemented Disc Regeneration in the Treatment of Patients With Low Back Pain With or Without Intervertebral Disc Herniation - VAST Trial
Brief Title: Viable Allograft Supplemented Disc Regeneration in the Treatment of Patients With Low Back Pain
Acronym: VAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VIVEX Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VAST - 001-017
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-04

CONDITIONS: Degenerative Disc Disease
Keywords: Chronic Lumbar Back Pain; Low Back Pain; Back Pain; Degenerative Disc Disease; Intervertebral Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain; Back Pain | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, randomized, parallel-arm study.
Who Masked: Participant
Masking Description: The assignment to treatment (active allograft, or placebo, or conservative care) is open label at Day 0 of the Active Phase to the extent that subjects receiving allograft or placebo will not be aware of what they have received, while those assigned to conservative care will be aware. All site study staff will be aware of the group to which each subject is randomized. Sites will be trained to ensure that subjects receiving the allograft or placebo treatment will remain blinded to their treatment throughout the study duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Allograft (Experimental): Injection of viable allograft
  Interventions: Other: Active Allograft
- Placebo (Placebo Comparator): Injection of saline
  Interventions: Other: Placebo
- Conservative Care (No Intervention): Continued conservative care treatment

INTERVENTIONS:
Other: Active Allograft — Injection of viable allograft into the nucleus pulposus of the degenerated disc
  Other Names: viable allograft disc injection; cellular allograft nucleus pulposus matrix
  Arms: Active Allograft
Other: Placebo — Injection of sterile normal saline (0.9% sodium chloride) into the nucleus pulposus of the degenerated disc
  Other Names: Saline injection; Placebo control
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of viable allograft transplantation for the treatment of patients with symptomatic disc degeneration and tissue loss.

All subjects randomized to Active Allograft will undergo injection of a viable allograft into the nucleus pulposus of the degenerated disc. All subjects randomized to Placebo will undergo injection with saline into the nucleus pulposus of the degenerated disc. All subjects randomized to Conservative Care will continue standard of care, with the opportunity to crossover at 3 months into the Active Allograft arm.

DETAILED DESCRIPTION:
This is a multicenter, prospective, parallel arm study to assess patients who participated in the VAST trial and receiving either viable allograft, saline, or allograft after cross-over. These patients will be evaluated at baseline, injection, 6 months, and 12 months. Subjects will then have an option for a 24 months and 36 months extension after their index procedures. Patients who received saline or active allograft in the VAST study will be allowed to receive viable allograft and followed for an additional 12 and 24 months after that election. These subjects will need to meet initial inclusion/exclusion criteria again before another injection.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide an English written Informed Consent
* Age 18 to 60 years inclusive
* Male or female
* Body mass index <35
* Pfirrmann Grade [3-6]
* Radiographic confirmation by MRI/X-ray of:

  1. translational instability defined as ≤5 mm, or
  2. angular instability defined as ≤5°
* Back pain (with or without radicular leg pain) measured by:

  1. ODI of at least 40%, and
  2. VASPI of at least 40mm
* Pathologic level between L1 and S1
* 1 or 2 vertebral level involvement that has been evaluated for at least 6 months and treated with conservative care
* Symptomatic back pain attributable to intervertebral disc for a minimum of 6 months
* No previous surgical treatment at the disc level(s) being considered
* Psychosocially, mentally and physically able to fully comply with this protocol, and follow-up schedule
* Ability to undergo allograft transplantation
* Life expectancy >2 years
* No contraindications to MRI
* No history of malignancy (basal cell carcinoma) or chronic infectious disease (e.g. HIV, Hepatitis)
* Agree to use appropriate contraception; not planning on becoming pregnant for 24 months after treatment
* Patient disc for transplant confirmed by inter-discal pressure measurement, or disc-imaging study.
* No signs or symptoms of infection
* No chronic use (>7 consecutive days) of anticoagulants (such as aspirin) or NSAIDs prior to treatment

Exclusion Criteria:

* Seropositive or seronegative spondyloarthropathy
* Type III Modic changes
* Prior surgeries of segments between L1 and S1
* Chemonucleolysis or percutaneous laserectomy of the affected disc prior to the study
* Chronic facet syndrome
* Stenosis of the spinal canal that is moderate to severe or more in degree
* Spondylodiscitis
* Spondylolisthesis (lysis and degenerative)
* Severe motor deficit or cauda equina disorder based on investigator determination
* Congenital abnormalities of the spinal nerves
* Pelvic and inguinal angiopathy
* Neurogenic inguinal syndrome
* Syringomyelia
* Diastematomyelia
* Traumatic neurological disorders
* Diseases of the kidney (nephritis, pyelonephritis)
* Other severe diseases of any other major body system as judged by the investigator
* Regular intake of systemic steroids
* Malignant diseases of any solid organ or any hematologic malignancy during the previous 5 years
* Patients who have participated in a clinical trial within the last month prior to inclusion
* Moderate to severe or greater lumbar stenosis of both transplantation endplates and adjacent levels

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 6 Months
  To evaluate the mean change from baseline in functional disability on the Oswestry Disability Index (ODI) measured from 0 (minimal disability) to 100 (maximal disability).
Oswestry Disability Index (ODI) | 12 Months
  To evaluate the mean change from baseline in functional disability on the Oswestry Disability Index (ODI) measured from 0 (minimal disability) to 100 (maximal disability).
Visual Analogue Scale of Pain Intensity (VASPI) | 6 Months
  To evaluate the mean change from baseline in chronic lumbar back pain scores on the Visual Analogue Scale of Pain Intensity (VASPI) measured from 0mm (no pain) to 100mm (worst pain).
Visual Analogue Scale of Pain Intensity (VASPI) | 12 Months
  To evaluate the mean change from baseline in chronic lumbar back pain scores on the Visual Analogue Scale of Pain Intensity (VASPI) measured from 0mm (no pain) to 100mm (worst pain).
Oswestry Disability Index (ODI) | 24 Months
  To evaluate the mean change from 12 months in functional durability on the Oswestry
Oswestry Disability Index (ODI) | 36 Months
  To evaluate the mean change from 12 months in functional durability on the Oswestry
Visual Analogue Scale of Pain Intensity (VASPI) | 24 Months
  To evaluate the mean change from 12 months in chronic lumbar back pain scores on the Visual Analogue Scale of Pain Intensity (VASPI) measured from 0mm (no pain) to 100mm (worst pain).
Visual Analogue Scale of Pain Intensity (VASPI) | 36 Months
  To evaluate the mean change from 12 months in chronic lumbar back pain scores on the Visual Analogue Scale of Pain Intensity (VASPI) measured from 0mm (no pain) to 100mm (worst pain).

SECONDARY OUTCOMES:
MRI Assessments | Baseline, 6 Months, and 12 Months
  To evaluate morphologic changes of treated intervertebral discs using MRI assessments.
X-Ray Assessments | Baseline, 6 Months, and 12 Months
  To evaluate morphologic changes of treated intervertebral discs using X-ray assessments.
36-Item Short Form Survey (SF-36) Questionnaire | Baseline, 6 Months, and 12 Months
  To evaluate results of the SF-36 Questionnaire.
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through study completion, an average of 12 months
  To evaluate the number of participants with treatment-related adverse events (AEs) and serious adverse events (SAEs).
Resource Utilization Questionnaire | Baseline, 6 Months, and 12 Months
  To evaluate results of the resource utilization questionnaire.
Oswestry Disability Index (ODI) | 6 and 12 Months
  To evaluate results of the ODI for improvement after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Ganey, PhD, Study Director — VIVEX Biologics, Inc.
Locations (13):
- United States (13):
  - Source Health, Santa Monica, California
  - IPM Medical Group, Walnut Creek, California
  - Laser Spine Institute, Tampa, Florida
  - Athens Orthopedic Clinic, Athens, Georgia
  - Neurological Institute of Savannah, Savannah, Georgia
  - OrthoIndy, Indianapolis, Indiana
  - Michigan Spine Clinic, Brownstown, Michigan
  - Ainsworth Institute of Pain Management, New York, New York
  - Clinical Investigations, LLC, Edmond, Oklahoma
  - Invictus Healthcare, Tulsa, Oklahoma
  - Texas Back Institute, Plano, Texas
  - Virginia iSpine Physicians, Richmond, Virginia
  - Gershon Pain Specialists, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hunter CW, Guyer R, Froimson M, DePalma MJ. Effect of age on outcomes after allogeneic disc tissue supplementation in patients with chronic discogenic low back pain in the VAST trial. Pain Manag. 2022 Apr;12(3):301-311. doi: 10.2217/pmt-2021-0078. Epub 2021 Dec 8. PMID 34875850
- [Derived] Beall DP, Davis T, DePalma MJ, Amirdelfan K, Yoon ES, Wilson GL, Bishop R, Tally WC, Gershon SL, Lorio MP, Meisel HJ, Langhorst M, Ganey T, Hunter CW. Viable Disc Tissue Allograft Supplementation; One- and Two-level Treatment of Degenerated Intervertebral Discs in Patients with Chronic Discogenic Low Back Pain: One Year Results of the VAST Randomized Controlled Trial. Pain Physician. 2021 Sep;24(6):465-477. No abstract available. PMID 34554689
- [Derived] Beall DP, Wilson GL, Bishop R, Tally W. VAST Clinical Trial: Safely Supplementing Tissue Lost to Degenerative Disc Disease. Int J Spine Surg. 2020 Apr 30;14(2):239-253. doi: 10.14444/7033. eCollection 2020 Apr. PMID 32355632

DOCUMENTS (2):
  • Study Protocol (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT03709901/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT03709901/SAP_001.pdf